CLINICAL TRIAL: NCT03632070
Title: A Study on Factors Related to Functional Recovery Using Brain Imaging of Stroke Patients
Brief Title: Factors Related to Functional Recovery Using Brain Imaging of Stroke Patients
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2018-07-168
Record Dates: First submitted 2018-08-13; First posted 2018-08-15 (Actual); Last update posted 2020-09-04 (Actual); Status verified 2020-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stroke: Patients with ischemic or hemorrhagic stroke who were admitted to Samsung Medical Center and transferred to the Department of Physical and Rehabilitation Medicine
  Interventions: Behavioral: Data acquisition of functional abilities

INTERVENTIONS:
Behavioral: Data acquisition of functional abilities — MRI data, motor evoked potentials, and behavior data acquisition

SUMMARY:
In this study, brain imaging predictive factors related to motor recovery will be investigated. Lastly, the prediction model will be established.

ELIGIBILITY:
Inclusion Criteria:

* Adults more than 19 years
* First-ever unilateral stroke
* Ischemic subacute stroke patients

Exclusion Criteria:

* Major active neurological disease or psychiatric disease
* Metallic implants in their brain
* Hemorrhagic stroke
* Bilateral lesions
* Recurrent stroke

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with ischemic stroke who were admitted to Samsung Medical Center and transferred to the Department of Physical and Rehabilitation Medicine
Sampling Method: Non-Probability Sample
Enrollment: 73 (Actual)
Dates: Start 2018-08-09 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment score at 3 months after stroke onset | 3 months after stroke onset]
  Measurement of motor function of upper and lower extremities

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No